CLINICAL TRIAL: NCT05091034
Title: The Efficacy of CAMP Air, a Web-based Asthma Intervention, Among Urban Adolescents With Uncontrolled Asthma
Brief Title: CAMP Air: Efficacy and Cost-effectiveness in Urban Adolescents
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: 3-C Institute for Social Development (Industry); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jean-Marie Bruzzese, Professor of Applied Developmental Psychology (in Nursing), Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAT2274; 1R61HL151958-01A1 (NIH)
Record Dates: First submitted 2021-10-12; First posted 2021-10-25 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Asthma
Keywords: Adolescents; E-Health; Intervention; Cost-effectiveness
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to 1 of 2 groups, an e-health intervention group or an education only control group.
Who Masked: Outcomes Assessor
Masking Description: The principal investigator responsible for evaluating the efficacy of the intervention and the research assistants conducting assessment interviews with adolescents and their caregiver will be blind to assigned arm conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAMP Air (Experimental): This is an e-health intervention consisting of 7 online modules. This behavioral intervention combines instruction, hands-on learning, interactive practice opportunities and tailored sessions. Teens learn about asthma, including treatment and triggers, the importance of seeing a medical provider and how they can overcome their specific barriers to seeing a medical provider, how they can talk to their parents about their asthma, and how they can care for their asthma, including managing stress and triggers. They also receive personalized feedback throughout the intervention and guidance on navigating the health care system.
  Interventions: Behavioral: Controlling Asthma Program for Adolescents (CAMP Air)
- Attention Control Asthma Education Intervention (Active Comparator): The control intervention consists of 7 online sessions delivered via PowerPoint slides with voice-over. Teens receive information on asthma and other related health conditions, such as stress and sleep, and will be given a list of relevant websites to learn more about these topics. They will learn how to monitor their health using checklists and will be referred to a medical provider for asthma and other conditions; if they do have a medical provider, they will be provided with a referral. The asthma education component for this group lacks the interactive and personalized elements of CAMP Air, differentiating it from the experimental arm.
  Interventions: Behavioral: Attention Control Asthma Education Intervention

INTERVENTIONS:
Behavioral: Controlling Asthma Program for Adolescents (CAMP Air) — Controlling Asthma Program for Adolescents (CAMP Air) is an e-health intervention grounded in social cognitive theory and motivational interviewing to guide teens through asthma self-care and how to navigate the health care system. It makes use of various interactive and personalized approaches.
  Other Names: CAMP Air
  Arms: CAMP Air
Behavioral: Attention Control Asthma Education Intervention — Using Asthma Plus, an asthma education program, teens learn about asthma and other conditions relevant to asthma and adolescents.
  Other Names: Asthma Plus
  Arms: Attention Control Asthma Education Intervention

SUMMARY:
This study will test the efficacy and cost-effectiveness of Controlling Asthma Program for Adolescents (CAMP Air), an e-health intervention, among urban predominately Black and Hispanic adolescents with uncontrolled asthma. It will also examine barriers and facilitators to adoption and implementation of CAMP Air in high-schools.

DETAILED DESCRIPTION:
Asthma prevalence and morbidity are high among adolescents, especially among Black and Hispanic youth. Yet, few interventions have been tested in adolescents. Despite the important role that technology plays in the lives of adolescents, only one intervention for adolescents with asthma is web-based. Additionally, research informing the scale-up of asthma interventions as well as their cost-effectiveness are scant. This study aims to address these treatment and methodological gaps by (1) systematically evaluating the efficacy of Controlling Asthma Program for Adolescents (CAMP Air), an e-health intervention, in urban adolescents with uncontrolled asthma; (2) assessing CAMP Air's cost-effectiveness; and (3) identifying multi-level factors associated with successful implementation of CAMP Air to inform its future scale-up. Due to COVID, at the start of the study, the spirometry data will not be collected from the participants (Secondary Outcomes 7 - 9).

The investigators plan to interview adolescents as the primary respondent for all outcomes.

Caregivers and school personnel are invited to be interviewed.

ELIGIBILITY:
Inclusion Criteria: Adolescents must report

* A prior diagnosis of asthma;
* Asthma medication use in the last 12 months; and
* Symptoms consistent with uncontrolled asthma, defined as: in the last month (a) daytime symptoms 3+ days a week, (b) night awakenings 3+ nights per month, or (c) activity limitations 3+ days per week; OR in the last 12 months (d) 2+ unscheduled visits to a clinic or medical provider because having asthma symptoms, (e) 2+ ED visits; (f) 1+ hospitalization for asthma, or (g) taken oral or systemic steroids in the past year.

Exclusion Criteria:

* Pregnant teenagers due to the stress of adolescent pregnancy and hormonal changes of pregnancy that could change asthma control;
* Students enrolled in 12th grade because those randomized to the control group will not be in the school the following school year to receive CAMP Air;
* Teenagers with a co-morbid disease or condition that might affect lung function, such as cystic fibrosis or sickle cell anemia; and
* Teenagers with highly specialized learning needs (e.g., Down's syndrome, mental retardation, severe ADHD) which may preclude completion of the intervention or assessments.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 374 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Mean score on the Asthma Control Questionnaire (ACQ-5) | Up to 1 year
  This measure, which is completed by the adolescents, assesses the adolescent's level of asthma control over the past week using 5-item version. The overall score is the mean of all questions; range = 0 - 6; lower scores indicate better control.
Total number of asthma-related urgent care visits | Up to 1 year
  This measure assesses the adolescent's number of asthma-related visits to a medical provider for urgent or immediate treatment, emergency room visits, and hospitalizations over 3 months. Completed by adolescents. Higher counts indicate more urgent health care utilization.

SECONDARY OUTCOMES:
Mean score on the Asthma Symptom Prevention Index | Up to 1 year
  This measure assesses the number of steps adolescents take to prevent the onset of symptoms. Completed by the adolescents. Score range = 0 - 9; higher scores indicate better asthma self-care.
Mean score on the Asthma Management Index | Up to 1 year
  This measure assesses the number of steps adolescents take to care for symptoms once they start. Completed by the adolescents. Score range = 0 - 7; higher scores indicate better asthma self-care.
Mean score on the Asthma Management Self-efficacy Index | Up to 1 year
  This measure assesses the confidence adolescents have in caring for their asthma. Completed by adolescents. Score range = 0 - 7; higher scores indicate better asthma management self-efficacy.
Proportion of adolescents taking controller medication | Up to 1 year
  Adolescents report the names of asthma medication they take, which will used to determine if controller medications are currently used.
Lung function - Overall functioning (Absolute ratio) | Up to 1 year
  The investigator will use spirometry to assess how well adolescents' lungs work. Spirometry is a test that measures how much air people can hold in their lungs as well as how much air they can exhale, or blow out, and how fast they can blow it out. The investigator will calculate the FEV1/FVC ratio, which is a proportion of how much air a person can exhale from the lung in the first second relative to the total amount of air that comes out during a full exhale. Forced expiratory volume (FEV) is the amount of air exhaled from the lung in one second and forced vital capacity (FVC) is the total amount of air that comes out during a full exhale. A ratio of 0.75 indicates the lungs are working well.
Lung Function - Obstruction to airflow (Maximum mid-expiratory flow rate) | Up to 1 year
  The investigators will use spirometry to assess how well air is flowing out of the smaller airways of the lungs via FEF25%-75%, or the maximum mid-expiratory flow rate. Forced expiratory flow (FEF) is the speed at which air comes out of the lungs during the middle portion of a person's full exhale. FEF25-75% is the average speed at which air flows out of the lungs from the moment a person has exhaled 25% of their full breathe to the moment they have exhaled 75% of their full breathe; it is expressed as a percentage. FEF25-75% values of more than 60% suggest normal airflow.
Lung function - Severity of impairment (FEV1% predicted) | Up to 1 year
  The investigators will use spirometry to assess how difficult it is for the adolescent's lungs to work when there is any indication that the lungs are not working properly. This will be measured as FEV1% predicted (FEV1% pred), and will be calculated by dividing the FEV1% of the adolescent by the average FEV1% in the population of adolescents with similar characteristics, such as age and sex. FEV1% is the FEV1/FVC absolute ratio expressed as a percentage. FEV1 is the amount of air exhaled from the lung in one second and FVC is the total amount of air that comes out during a full exhale. FEV1% pred values of 69 or less indicate moderate to severe difficulties in lung functioning; values of 70 or greater indicate mild difficulties in lung functioning.
Mean score on the Paediatric Asthma Quality of Life Questionnaire | Up to 1 year
  Adolescents complete the Paediatric Asthma Quality of Life Questionnaire, which measures how they have felt in the past week because of their asthma. Comprised of 3 sub scales, which are combined for an overall mean score ranging from 1 - 7; higher scores indicate better pediatric asthma quality of life.
Total number of oral steroid bursts | Up to 1 year
  Using the list of medications obtained from adolescents, the investigator will determine if there is use of oral steroids. If so, adolescents will also be asked how many times those medications were used over a period of 5 to 7 days in 3 months. Oral steroids are medications used to reduce acute inflammation and swelling in the lungs when other asthma medications are not working. A burst refers to a single period of 5 to 7 days in which a person takes oral steroids.
Total number of days with asthma symptoms | Up to 1 year
  Adolescents report the number of days they had asthma symptoms over the last 2 weeks.
Total number of nights woken due to asthma | Up to 1 year
  Adolescents report on how many nights asthma symptoms disrupted sleep or caused wakening over 2 weeks.
Total number of days with activity limitations due to asthma | Up to 1 year
  Adolescents report on the number of days usual activities could not be carried out over 2 weeks due to asthma.
Total number of school absences due to asthma | Up to 1 year
  Adolescents report on the number of days school was missed due to asthma over 2 weeks.
Frequency of school absences due to asthma | Up to 1 year
  Adolescents reporting any school absences due to asthma in the last 2 weeks will also be asked how typical this attendance was over 3 months.
Total number of school absences | Up to 1 year
  The investigators will compute adolescents' total number of school absences, regardless of the reason, from attendance records obtained from each school.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marie Bruzzese, PhD, Principal Investigator — Columbia University
Locations (1):
- High schools in the 5 boroughs of New York City, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The 3-C Institute will house the web-based intervention on their server, and conduct all data management activities for the study. Data stored electronically and shared between sites will be de-identified by HIPAA standards using the "safe-harbor" method (i.e., all 18 identifiers will be stripped) whenever possible, otherwise it will be sent encrypted. Data will be stored on a password-protected webserver.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Up to 7 years from the end of the study
Access Criteria: De-identified

REFERENCES:
- [Background] Zahran HS, Bailey CM, Damon SA, Garbe PL, Breysse PN. Vital Signs: Asthma in Children - United States, 2001-2016. MMWR Morb Mortal Wkly Rep. 2018 Feb 9;67(5):149-155. doi: 10.15585/mmwr.mm6705e1. PMID 29420459
- [Background] Glick AF, Tomopoulos S, Fierman AH, Trasande L. Disparities in Mortality and Morbidity in Pediatric Asthma Hospitalizations, 2007 to 2011. Acad Pediatr. 2016 Jul;16(5):430-437. doi: 10.1016/j.acap.2015.12.014. Epub 2016 Jan 6. PMID 26768727
- [Background] Sullivan P, Ghushchyan VG, Navaratnam P, Friedman HS, Kavati A, Ortiz B, Lanier B. School absence and productivity outcomes associated with childhood asthma in the USA. J Asthma. 2018 Feb;55(2):161-168. doi: 10.1080/02770903.2017.1313273. Epub 2017 Apr 28. PMID 28453370
- [Background] Pearlman DN, Zierler S, Meersman S, Kim HK, Viner-Brown SI, Caron C. Race disparities in childhood asthma: does where you live matter? J Natl Med Assoc. 2006 Feb;98(2):239-47. PMID 16708510
- [Background] Akinbami LJ, Moorman JE, Garbe PL, Sondik EJ. Status of childhood asthma in the United States, 1980-2007. Pediatrics. 2009 Mar;123 Suppl 3:S131-45. doi: 10.1542/peds.2008-2233C. PMID 19221156
- [Background] Park E, Kwon M. Health-Related Internet Use by Children and Adolescents: Systematic Review. J Med Internet Res. 2018 Apr 3;20(4):e120. doi: 10.2196/jmir.7731. PMID 29615385
- [Background] Bruzzese JM, Sheares BJ, Vincent EJ, Du Y, Sadeghi H, Levison MJ, Mellins RB, Evans D. Effects of a school-based intervention for urban adolescents with asthma. A controlled trial. Am J Respir Crit Care Med. 2011 Apr 15;183(8):998-1006. doi: 10.1164/rccm.201003-0429OC. Epub 2010 Dec 7. PMID 21139088
- [Background] Joseph CL, Peterson E, Havstad S, Johnson CC, Hoerauf S, Stringer S, Gibson-Scipio W, Ownby DR, Elston-Lafata J, Pallonen U, Strecher V; Asthma in Adolescents Research Team. A web-based, tailored asthma management program for urban African-American high school students. Am J Respir Crit Care Med. 2007 May 1;175(9):888-95. doi: 10.1164/rccm.200608-1244OC. Epub 2007 Feb 8. PMID 17290041
- [Background] Hollenbach JP, Cloutier MM. Implementing school asthma programs: Lessons learned and recommendations. J Allergy Clin Immunol. 2014 Dec;134(6):1245-1249. doi: 10.1016/j.jaci.2014.10.014. PMID 25482869
- [Background] Koh S, Lee M, Brotzman LE, Shelton RC. An orientation for new researchers to key domains, processes, and resources in implementation science. Transl Behav Med. 2020 Feb 3;10(1):179-185. doi: 10.1093/tbm/iby095. PMID 30445445
- [Background] Brownson RC, Colditz GA, Proctor EK. Dissemination and Implementation Research in Health: Translating Science to Practice (2nd Edition). New York: Oxford University Press; 2018.
- [Background] Bruzzese JM, George M, Liu J, Evans D, Naar S, DeRosier ME, Thomas JM. The Development and Preliminary Impact of CAMP Air: A Web-based Asthma Intervention to Improve Asthma Among Adolescents. Patient Educ Couns. 2021 Apr;104(4):865-870. doi: 10.1016/j.pec.2020.09.011. Epub 2020 Sep 15. PMID 33004234